CLINICAL TRIAL: NCT01084252
Title: A Phase I/2 Dose Escalation Safety, Pharmacokinetic and Efficacy Study of Multiple Intravenous Administrations of a Humanized Monoclonal Antibody (SAR650984) Against CD38 in Patients With Selected CD38+ Hematological Malignancies
Brief Title: Phase 1/2 Dose Escalation and Efficacy Study of Anti-CD38 Monoclonal Antibody in Patients With Selected CD38+ Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED10893; U1111-1116-5472 (Registry Identifier: ICTRP); 2013-001418-13 (EudraCT Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Hematological Malignancy
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Hematologic Neoplasms | interventions — isatuximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (14):
- Phase 1:Isatuximab <=1 mg/kg Q2W (Experimental): Participants with CD38+ hematological malignancies (HM), received Isatuximab at any one of the dose less than or equal to (<=) 1 milligram per kilogram (mg/kg) (i.e. either 0.0001 mg/kg or 0.001 mg/kg or 0.01 mg/kg or 0.03 mg/kg or 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg) as intravenous (IV) infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1: Isatuximab 3mg/kg Q2W (Experimental): Participants with CD38+ HM, received Isatuximab 3 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1: Isatuximab 5 mg/kg Q2W (Experimental): Participants with CD38+ HM, received Isatuximab 5 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) (Experimental): Participants with CD38+ HM along with participants with standard risk multiple myeloma were included this arm and, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1:Isatuximab (CD38 + HM and High Risk Multiple Myeloma) (Experimental): Participants with CD38+ HM along with participants with high risk multiple myeloma, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1: Isatuximab 10 mg/kg QW (Experimental): Participants with CD38+ HM, received Isatuximab 10 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1: Isatuximab 20 mg/kg Q2W (Experimental): Participants with CD38+ HM, received Isatuximab 20 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 1: Isatuximab 20 mg/kg QW (Experimental): Participants with CD38+ HM, received Isatuximab 20 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W (Experimental): Participants with multiple Myeloma received Isatuximab 3 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable adverse event (AE), disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Stage 1a: Isatuximab 10 mg/kg Q2W (Experimental): Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase2 Stage1a:Isatuximab 10mg/kg Q2W; Then Q4W (Experimental): Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion Q2W, i.e. on Day 1 and Day 15 of Cycle 1 and 2 (each cycle 28 days), then every 4 week (Q4W), i.e. on Day 1 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W (Experimental): Participants with multiple Myeloma received Isatuximab 20 mg/kg, as IV infusion QW, i.e. on Day 1, 8, 15 and 22 of Cycle 1 and 2 (each cycle 28 days), then Q2W, i.e. on Day 1 and Day 15 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 92 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Stage 2: Isatuximab Alone (Experimental): Participants with relapsed or relapsed/refractory multiple myeloma (RRMM), received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 301 weeks).
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Stage 2: Isatuximab + Dexamethasone (Experimental): Participants with relapsed or RRMM, received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles along with dexamethasone: tablet or as IV infusion (40 mg/day for less than [<] 75 years of age; 20 mg/day [greater than or equal to [>=] for 75 years of age) on Days 1, 8, 15 and 22 of each 28 days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 301 weeks).
  Interventions: Drug: Isatuximab SAR650984; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: Dexamethasone — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Arms: Phase 2 Stage 2: Isatuximab + Dexamethasone
Drug: Dexamethasone — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Phase 2 Stage 2: Isatuximab + Dexamethasone

SUMMARY:
Primary Objective:

Phase 1:

To determine the maximum tolerated dose (MTD)/maximum administered dose (MAD) of SAR650984 (Isatuximab).

Phase 2 (stage 1):

To evaluate the activity of single-agent Isatuximab at different doses/schedules and to select dose and regimen to further evaluate the overall response rate (ORR) of Isatuximab as single agent or in combination with dexamethasone.

Phase 2 (stage 2):

To evaluate the activity in terms of overall response rate (ORR) of Isatuximab at the selected dose/schedule from stage1, as single agent (ISA arm) and in combination with dexamethasone (ISAdex arm).

Secondary Objectives:

Phase 1:

* To characterize the global safety profile including cumulative toxicities.
* To evaluate the pharmacokinetic (PK) profile of Isatuximab in the proposed dosing schedule(s).
* To assess the pharmacodynamics (PD), immune response, and preliminary disease response.

Phase 2 (stage 1): to evaluate the following objectives for Isatuximab as single agent:

* Safety
* Efficacy as measured by duration of response, clinical benefit rate, progression free survival, overall survival.

Phase 2 (stage 2): to evaluate the following objectives in each arm (ISA and ISAdex):

* Safety
* Efficacy as measured by duration of response, clinical benefit rate, progression free survival, overall survival.
* Participant-reported changes in health-related quality of life, symptoms of multiple myeloma and generic health status.
* Pharmacokinetic profile of Isatuximab.
* Immunogenicity of Isatuximab.
* Investigate the relationship between CD38 receptor density and CD38 receptor occupancy (Stage 1 only) on multiple myeloma cells and parameters of clinical response.

DETAILED DESCRIPTION:
The Phase 1 study duration for an individual participant included a screening period for inclusion of up to 2 weeks, treatment with Isatuximab QW (every week) or Q2W (every 2 weeks) unless discontinued earlier due to safety or disease progression. Participants were followed for a minimum of 30 days following the last use of study drug or more than 30 days in case of unresolved toxicity, or up to initiation of another anticancer treatment.

The Phase 2 study duration for an individual participant included a screening period for inclusion of up to 3 weeks, then a treatment period and a follow up period. Treatment was continued until disease progression, unacceptable adverse reactions or other reasons for discontinuation. Participants were followed every 3 months following the last use of study drug until death or study cutoff, whichever came first.

ELIGIBILITY:
Inclusion criteria:

Phase 1:

* For dose escalation cohorts, participants with confirmed selected CD38+ hematological malignancies as specified below who had progressed on after standard therapy or for whom there was no effective standard therapy (refractory/relapsed participants). B-cell Non-Hodgkin-lymphoma/leukemia (NHL) participants with at least 1 measurable lesion. Multiple myeloma (MM) participants with measurable M-protein serum and/or 24-hour urine. Acute myeloid leukemia (AML) participants, all types except M3 based on French-American-British (FAB) classification. Acute Lymphoblastic Leukemia (B-cell ALL) participants. Chronic lymphocytic leukemia (CLL) participants.
* For expansion cohorts, participants with relapsed/refractory MM with measurable M-protein (serum M-protein of >0.5 g/dL and/or urine M-protein of >200 mg (24-hr urine)) or elevated serum free light chains (FLC) >10 mg/dL with abnormal FLC ratio) who had progressed on or after standard therapy that included an Immunomodulatory drug (IMiD) and a proteasome inhibitor and who met the protocol defined criteria for standard risk or high risk.

Phase 2:

* Participants had a known diagnosis of multiple myeloma with evidence of measurable disease, and have evidence of disease progression based on International Myeloma Working Group (IMWG) criteria: Serum M-protein ≥1 g/dL, or urine M-protein >=200 mg/24 hours or in the absence of measurable m-protein, serum FLC >=10 mg/dL, and abnormal serum immunoglobulin kappa lambda FLC ratio (<0.26 or >1.65).
* Participants who received at least three prior lines of therapy for MM and had treatment with an IMiD (for >=2 cycles or >=2 months of treatment) and a proteasome inhibitor (PI) (for >=2 cycles or >=2 months of treatment) OR participants whose disease was double refractory to an IMiD and a PI. For participants who had received more than 1 type of IMiD and PI, their disease must be refractory to the most recent one.
* Participants who had achieved a minimal response or better to at least one prior line of therapy.
* Participants who had received an alkylating agent (>=2 cycles or >=2 months) either alone or in combination with other MM treatments.
* Stage 2 only: Participants who had evidence of disease progression on or after the most recent prior regimen based on IMWG criteria.

Exclusion criteria:

Phase 1:

* Karnofsky performance status <60
* Poor bone marrow reserve
* Poor organ function
* Known intolerance to infused protein products, sucrose, histidine, polysorbate 80 or known hypersensitivity to any of the components of the study therapy that was not amenable to pre-medication with steroids and H2 blockers
* Any serious active disease (including clinically significant infection that was chronic, recurrent, or active) or co-morbid condition, which, in the opinion of the investigator, interfered with the safety, the compliance with the study or with the interpretation of the results
* Any severe underlying medical conditions including presence of laboratory abnormalities, which could impair the ability to participate in the study or the interpretation of its results

Phase 2:

* Participants with multiple myeloma immunoglobulin M (IgM) subtype
* Previous treatment with any anti-CD38 therapy
* Participants with concurrent plasma cell leukemia
* Participants with known or suspected amyloidosis
* Karnofsky performance status <60 (stage 1)/Eastern Cooperative Oncology Group (ECOG) Performance status >2 (stage 2).
* Poor bone marrow reserve
* Poor organ function
* Known intolerance to infused protein products, sucrose, histidine, polysorbate 80 or known hypersensitivity to any of the components of the study therapy that was not amenable to pre-medication with steroids and H2 blockers
* Any serious active disease (including clinically significant infection that was chronic, recurrent, or active) or co-morbid condition, which, in the opinion of the investigator, interfered with the safety, the compliance with the study or with the interpretation of the results
* Any severe underlying medical conditions including presence of laboratory abnormalities, which impaired the ability to participate in the study or the interpretation of its results

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (59):
- United States (16):
  - Mayo Clinic Site Number : 840003, Scottsdale, Arizona
  - UCSF MS Center Site Number : 840005, San Francisco, California
  - Emory University Site Number : 840009, Atlanta, Georgia
  - University of Chicago Site Number : 840010, Chicago, Illinois
  - The University Of Michigan Site Number : 840022, Ann Arbor, Michigan
  - Karmanos Cancer Center Site Number : 840027, Detroit, Michigan
  - Mayo Clinic of Rochester Site Number : 840018, Rochester, Minnesota
  - Washington University School of Medicine Site Number : 840013, St Louis, Missouri
  - The Cancer Center At Hackensack University Medical Site Number : 840011, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center Site Number : 840014, New York, New York
  - Duke University Medical College Site Number : 840016, Durham, North Carolina
  - University of Cincinnati Site Number : 840004, Cincinnati, Ohio
  - Vanderbilt University Site Number : 840001, Nashville, Tennessee
  - Huntsman Cancer Institute at the University of Utah Site Number : 840002, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center Site Number : 840012, Seattle, Washington
  - Medical College of Wisconsin Site Number : 840017, Milwaukee, Wisconsin
- Argentina (3):
  - Investigational Site Number : 032003, Capital Federal, Buenos Aires
  - Investigational Site Number : 032002, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Investigational Site Number : 032001, Ciudad de Buenos Aires, Buenos Aires
- Investigational Site Number : 056001, Antwerp, Belgium
- Brazil (4):
  - Hospital Mae de Deus Site Number : 076003, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor - Hospital do Cancer de Barretos - Fundacao Pio XII Site Number : 076001, Barretos, São Paulo
  - Clínica São Germano Site Number : 076002, São Paulo, São Paulo
  - Instituto COI de Educacao e Pesquisa Site Number : 076004, Rio de Janeiro
- Investigational Site Number : 152001, Temuco, La Araucanía, Chile
- Finland (2):
  - Investigational Site Number : 246001, Helsinki
  - Investigational Site Number : 246002, Turku
- France (3):
  - Investigational Site Number : 250003, Nantes
  - Investigational Site Number : 250004, Pierre-Bénite
  - Investigational Site Number : 250001, Toulouse
- Investigational Site Number : 300001, Athens, Greece
- Israel (2):
  - Investigational Site Number : 376004, Jerusalem
  - Investigational Site Number : 376002, Tel Litwinsky
- Italy (2):
  - Investigational Site Number : 380001, Bologna
  - Investigational Site Number : 380002, Torino
- Mexico (2):
  - Investigational Site Number : 484003, San Luis Potosí City, San Luis Potosí
  - Investigational Site Number : 484001, Monterrey
- Peru (2):
  - Investigational Site Number : 604001, Arequipa
  - Investigational Site Number : 604002, Lima
- Russia (4):
  - Investigational Site Number : 643002, Moscow
  - Investigational Site Number : 643003, Novosibirsk
  - Investigational Site Number : 643001, Petrozavodsk
  - Investigational Site Number : 643004, Saint Petersburg
- Spain (7):
  - Investigational Site Number : 724005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 724007, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 724002, Pamplona, Navarre
  - Investigational Site Number : 724006, Valencia, Valenciana, Comunidad
  - Investigational Site Number : 724004, Madrid
  - Investigational Site Number : 724001, Salamanca
  - Investigational Site Number : 724008, Seville
- Turkey (Türkiye) (4):
  - Investigational Site Number : 792002, Ankara
  - Investigational Site Number : 792005, Ankara
  - Investigational Site Number : 792001, Istanbul
  - Investigational Site Number : 792004, Samsun
- Ukraine (3):
  - Investigational Site Number : 804001, Kyiv
  - Investigational Site Number : 804004, Vinnytsia
  - Investigational Site Number : 804002, Zaporizhzhya
- United Kingdom (2):
  - Investigational Site Number : 826002, Southampton, Hampshire
  - Investigational Site Number : 826001, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dimopoulos M, Bringhen S, Anttila P, Capra M, Cavo M, Cole C, Gasparetto C, Hungria V, Jenner M, Vorobyev V, Ruiz EY, Yin JY, Saleem R, Hellet M, Mace S, Paiva B, Vij R. Isatuximab as monotherapy and combined with dexamethasone in patients with relapsed/refractory multiple myeloma. Blood. 2021 Mar 4;137(9):1154-1165. doi: 10.1182/blood.2020008209. PMID 33080623
- [Derived] Mikhael J, Richter J, Vij R, Cole C, Zonder J, Kaufman JL, Bensinger W, Dimopoulos M, Lendvai N, Hari P, Ocio EM, Gasparetto C, Kumar S, Oprea C, Chiron M, Brillac C, Charpentier E, San-Miguel J, Martin T. A dose-finding Phase 2 study of single agent isatuximab (anti-CD38 mAb) in relapsed/refractory multiple myeloma. Leukemia. 2020 Dec;34(12):3298-3309. doi: 10.1038/s41375-020-0857-2. Epub 2020 May 14. PMID 32409691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were involved in the study from 11 May 2010 at 59 centers in 18 countries. A total of 418 participants were screened, of which 351 participants were enrolled. A total of 67 participants had screen failures due to failure to meet inclusion criteria.
Pre-assignment Details: Study consisted 2 phases: Phase 1 and Phase 2. Phase 1 was a dose escalation part of isatuximab to determine maximum tolerated dose (MTD). Phase 2 was conducted for efficacy and safety evaluation of isatuximab with or without dexamethasone. It consisted of 2 stages: Stage 1 (comprised of 1a and 1b) and Stage 2.
Groups:
- Phase1: Isatuximab <=1 mg/kg Every 2 Weeks (Q2W): Participants with CD38+ hematological malignancies (HM), received Isatuximab at any one of the dose less than or equal to (<=) 1 milligram per kilogram (mg/kg) (i.e. either 0.0001 mg/kg or 0.001 mg/kg or 0.01 mg/kg or 0.03 mg/kg, or 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg) as intravenous (IV) infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma): Participants with CD38+ HM along with participants with standard risk multiple myeloma were included in this arm and, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma): Participants with CD38+ HM along with participants with high risk multiple myeloma were included in this arm and, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 10 mg/kg Every Week (QW): Participants with CD38+ HM, received Isatuximab 10 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W: Participants with multiple Myeloma received Isatuximab 3 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion Q2W, i.e. on Day 1 and Day 15 of Cycle 1 and 2 (each cycle 28 days), then every 4 weeks (Q4W), i.e. on Day 1 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
- Phase 2 Stage 2: Isatuximab + Dexamethasone: Participants with relapsed or RRMM, received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles along with dexamethasone: tablet or as IV infusion (40 mg/day for less than [<] 75 years of age; 20 mg/day for greater than or equal to [>=] 75 years of age) on Days 1, 8, 15 and 22 of each 28 days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 301 weeks).
Period: Phase 1 (120 Weeks)
Arm/Group | Phase1: Isatuximab <=1 mg/kg Every 2 Weeks (Q2W) | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5 mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg Every Week (QW) | Phase 1: Isatuximab 20 mg/kg Q2W | Phase 1: Isatuximab 20 mg/kg QW | Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Started | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
All Treated (AT) Population (Participants who signed informed consent & received at least 1 dose/even incomplete of isatuximab.) | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Participants with end of treatment or death from any cause forms completed.) | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Stage 1(1a-414Weeks;1b-92Weeks)
Arm/Group | Phase1: Isatuximab <=1 mg/kg Every 2 Weeks (Q2W) | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5 mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg Every Week (QW) | Phase 1: Isatuximab 20 mg/kg Q2W | Phase 1: Isatuximab 20 mg/kg QW | Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.) | 24 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.) | 25 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.) | 25 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.) | 0 | 0
AT Population (Participants who signed informed consent & received at least 1 dose/even incomplete of isatuximab.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 24 | 25 | 25 | 0 | 0
Completed (Participants with end of treatment or death from any cause forms completed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 24 | 25 | 25 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Stage 2 (301 Weeks)
Arm/Group | Phase1: Isatuximab <=1 mg/kg Every 2 Weeks (Q2W) | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5 mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg Every Week (QW) | Phase 1: Isatuximab 20 mg/kg Q2W | Phase 1: Isatuximab 20 mg/kg QW | Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 110 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.) | 55 (Phase 1, Phase 2 Stage 1 and Phase 2 Stage 2 were separate populations.)
AT Population (Participants who signed informed consent & received at least 1 dose/even incomplete of isatuximab.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 109 | 55
Completed (Participants with end of treatment or death from any cause forms completed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 109 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Enrolled, but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on AT population.
Groups:
- Phase 1:Isatuximab <=1 mg/kg Q2W: Participants with CD38+ HM, received Isatuximab at any one of the dose <= 1 mg/kg (i.e. either 0.0001 mg/kg or 0.001 mg/kg or 0.01 mg/kg or 0.03 mg/kg, or 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg) as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Total: Total of all reporting groups
Arm/Group | Phase 1:Isatuximab <=1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5 mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg QW | Phase 1: Isatuximab 20 mg/kg Q2W | Phase 1: Isatuximab 20 mg/kg QW | Phase 2 Stage 1a: Isatuximab 3 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10 mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone | Total
Number analyzed (Participants) | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7 | 23 | 24 | 25 | 25 | 109 | 55 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.6) | 63.5 (6.2) | 62.0 (3.5) | 65.0 (7.2) | 60.8 (12.6) | 61.7 (12.7) | 63.3 (10.0) | 60.0 (8.3) | 63.2 (8.9) | 63.9 (8.8) | 61.0 (7.3) | 61.1 (10.3) | 66.6 (8.8) | 66.3 (8.9) | 64.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 1 | 11 | 9 | 2 | 2 | 3 | 11 | 11 | 7 | 13 | 58 | 26 | 162
  Male | 11 | 3 | 2 | 15 | 9 | 4 | 5 | 4 | 12 | 13 | 18 | 12 | 51 | 29 | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 3 | 5 | 3 | 20
  White | 14 | 4 | 3 | 20 | 13 | 4 | 6 | 7 | 21 | 19 | 19 | 21 | 91 | 45 | 287
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 6 | 2 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 11 | 6 | 35

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were assessed using the national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 4.03. DLTs were defined as any Grade 3 or higher non-hematological toxicity (with the exception of allergic reaction/hypersensitivity), Grade 4 neutropenia and/or Grade 4 thrombocytopenia lasting longer than 5 days, attributed to isatuximab. Any other toxicity that the Investigator and the Sponsor deemed to be dose-limiting, regardless of the grade, was also considered as DLT.
Time Frame: Day 1 of Cycle 1 up to Day 14 of Cycle 2
Population: DLT evaluable population included participants who gave their informed consent, received at least 1 dose of isatuximab during Phase 1 and had a DLT assessment at the end of Cycle 2. Data was planned not to be collected and analyzed for the arm: Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Isatuximab 5mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 5 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 20mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 20 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 20mg/kg QW: Participants with CD38+ HM, received Isatuximab 20 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of DLT, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1:Isatuximab <=1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 14 | 6 | 3 | 6 | 6 | 6 | 6
Participants | 1 | 1 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. TEAEs were defined as AEs that developed or worsened during the on-treatment period which was defined as the period from the time of first dose of study treatment until 30 days after the last dose of study treatment.
Time Frame: From Baseline up to 30 days after the last dose (maximum duration: 120 weeks )
Population: Analysis was performed on AT population which included participants who signed informed consent and received at least 1 dose/even incomplete of isatuximab.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Isatuximab <=1mg/kg Q2W: Participants with CD38+ HM, received Isatuximab at any one of the dose <= 1 mg/kg (i.e. either 0.0001 mg/kg or 0.001 mg/kg or 0.01 mg/kg or 0.03 mg/kg, or 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg) as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1: Isatuximab <=1mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7
Participants | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 6

3. Primary Outcome: Phase 2 Stage 1: Percentage of Participants With Overall Response (OR) According to International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: OR defined as participants with stringent complete response (sCR) or complete response (CR) or very good partial response (VGPR) or partial response (PR) . Based on IMWG, CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow; sCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; PR: >=50% reduction of serum M-Protein and reduction in urinary M-protein by >=90% or to <200 mg/24 hours; >=50% decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria or a >=50% reduction in plasma cells in place of M-protein if present at baseline.
Time Frame: From the date of randomization until disease progression or death or data cut-off (maximum duration: 77 weeks for Stage 1a arms and 53 weeks for Stage 1b arm)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 Stage 1a: Isatuximab 3 mg/kg: Participants with multiple Myeloma received Isatuximab 3 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
- Phase 2 Stage 1a: Isatuximab 10 mg/kg: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W and Then Q4W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion Q2W, i.e. on Day 1 and Day 15 of Cycle 1 and 2 (each cycle 28 days), then Q4W, i.e. on Day 1 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
- Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W: Participants with multiple Myeloma received Isatuximab 20 mg/kg, as IV infusion QW, i.e. on Day 1, 8, 15 and 22 of Cycle 1 and 2 (each cycle 28 days), then Q2W, i.e. on Day 1 and Day 15 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 53 weeks).
Arm/Group | Phase 2 Stage 1a: Isatuximab 3 mg/kg | Phase 2 Stage 1a: Isatuximab 10 mg/kg | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W and Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 23 | 24 | 25 | 25
percentage of participants | 4.3 | 29.2 | 20.0 | 24.0

4. Primary Outcome: Phase 2 Stage 2: Percentage of Participants With Overall Response According to Updated IMWG Response Criteria
Description: OR: participants with sCR or CR or VGPR or PR. As per updated IMWG, CR: Negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow; normal FLC ratio of 0.26-1.65 in participants with only FLC disease; sCR: CR and normal FLC ratio and no clonal cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours, >90% decrease in the difference between involved and uninvolved FLC levels; PR: >=50% reduction of serum M-Protein and reduction in urinary M-protein by >=90% or to <200 mg/24 hours; >=50% decrease in the difference between involved and uninvolved FLC levels in place of M-protein criteria or >=50% reduction in plasma cells in place of M-protein if present at baseline.
Time Frame: From the date of randomization to date of death from any cause (maximum duration: 97 weeks)
Population: Analysis was performed on AT population which included participants who signed informed consent & received at least 1 dose/even incomplete of isatuximab.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 Stage 2: Isatuximab Alone: Participants with relapsed or relapsed/refractory multiple myeloma (RRMM), received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 97 weeks).
- Phase 2 Stage 2: Isatuximab + Dexamethasone: Participants with relapsed or RRMM, received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles along with dexamethasone: tablet or as IV infusion (40 mg/day for less than [<] 75 years of age; 20 mg/day for greater than or equal to [>=] 75 years of age) on Days 1, 8, 15 and 22 of each 28 days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 97 weeks).
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 109 | 55
percentage of participants | 23.9 | 43.6

5. Secondary Outcome: Pharmacokinetic (PK) Assessment: Phase 1: Plasma Concentration of Isatuximab Observed at the End of an Intravenous Infusion (Ceoi)
Description: Ceoi was defined as the plasma concentration of Isatuximab at end of infusion. Data for this outcome measure was planned to be collected and analyzed separately for dose 0.3 mg/kg, 1 mg/kg and not for 0.0001, 0.001, 0.01, 0.03 and 0.1 dose levels (reported under one arm, i.e. Phase 1: Isatuximab <=1mg/kg in participant flow). Analysis was performed on PK population: participants who gave informed consent, received at least one dose (even if incomplete) of isatuximab, had an assessable PK parameter.
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1: At the end of infusion
Population: Here, "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure and "0" in "number analyzed" field signifies none of the participant were evaluable because at Cycle 3, Day 1, only data for reporting arms "Phase 1: Isatuximab 10mg/kg QW" and "Phase 1: Isatuximab 20mg/kg QW" was planned to be collected and analyzed.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Groups:
- Phase 1: Isatuximab 0.3 mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 0.3 mg/kg, as IV infusion on Day 1of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 1 mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 1 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 10mg/kg QW: Participants with CD38+ HM, received Isatuximab 10 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of unaccepted toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1: Isatuximab 0.3 mg/kg Q2W | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 6 | 3 | 4 | 2 | 15 | 5 | 3 | 4 | 6
microgram per milliliter (mcg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 3 | 4 | 2 | 15 | 5 | 3 | 3 | 6
  Cycle 1 Day 1 | 2.08667 (0.65567) | 13.18333 (5.74464) | 44.22500 (15.30651) | 125.50000 (53.03301) | 171.43333 (50.18853) | 148.80000 (18.48513) | 400.33333 (52.51984) | 173.33333 (20.64784) | 334.33333 (98.28462)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
  Cycle 3 Day 1 |  |  |  |  |  |  |  | 299.82500 (220.83898) | 715.33333 (188.01241)

6. Secondary Outcome: PK Assessment: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Isatuximab
Description: Data for this outcome measure was planned to be collected and analyzed separately for dose 0.3 mg/kg, 1 mg/kg and not for 0.0001, 0.001, 0.01, 0.03 and 0.1 dose levels (reported under one arm, i.e. Phase 1: Isatuximab <=1mg/kg in participant flow). Analysis was performed on PK population.
Time Frame: For Q2W:Cycle 1,Day 1: pre-dose, 15 min after start of infusion, at the end of infusion, 3, 7, 24, 48 and 168 hr post-infusion; For QW: Cycle 1,Day 1: pre-dose, 15 min after start of infusion, at the end of infusion, 4, 24, 48, 72 and 168 hr post-infusion
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Phase 1: Isatuximab 0.3 mg/kg Q2W | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 6 | 3 | 4 | 2 | 11 | 5 | 3 | 4 | 6
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 3 | 4 | 2 | 11 | 5 | 3 | 3 | 6
  Cycle 1 Day 1 | 2.00 (31) | 12.4 (45) | 53.7 (28) | 126 (NA) — Geometric Coefficient of Variation was not calculated because it was pre-specified not to calculate the value if number of participants was <=2. | 181 (48) | 154 (13) | 457 (28) | 181 (20) | 343 (29)
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
  Cycle 3 Day 1 |  |  |  |  |  |  |  | 265 (67) | 712 (27)

7. Secondary Outcome: PK Assessment: Phase 1: Time to Reach Maximum Plasma Concentration Observed (Tmax) of Isatuximab
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Isatuximab 0.3 mg/kg Q2W | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 6 | 3 | 4 | 2 | 11 | 5 | 3 | 4 | 6
hours
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 3 | 4 | 2 | 11 | 5 | 3 | 3 | 6
  Cycle 1 Day 1 | 2.49 [1.42 to 3.43] | 4.35 [3.13 to 6.33] | 6.99 [4.58 to 8.00] | 7.65 [5.13 to 10.17] | 4.28 [2.15 to 9.37] | 4.92 [2.60 to 30.08] | 5.87 [5.78 to 9.90] | 2.25 [2.20 to 7.50] | 6.83 [3.98 to 10.53]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
  Cycle 3 Day 1 |  |  |  |  |  |  |  | 4.30 [2.57 to 27.48] | 8.07 [2.87 to 29.03]

8. Secondary Outcome: PK Assessment: Phase 1: Plasma Concentration of Isatuximab at Week 1, 2 and 3
Description: Data for this outcome measure was planned to be collected and analyzed only for dose 1 mg/kg and not for 0.0001, 0.001, 0.01, 0.03, 0.1 and 0.3 mg/kg dose levels (reported under one arm, i.e. Phase 1: Isatuximab <=1mg/kg in participant flow).
Time Frame: Week 1, 2 and 3
Population: Analysis was performed on PK population. Here, 'number analyzed' = number of participants with available data for each category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Phase 1: 5mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 5 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10 mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 3 | 6 | 3 | 18 | 16 | 6 | 6 | 7
mcg/mL
  Week 1 | 0.00223 (86) | 1.44 (85) | 15.3 (90) | 27.6 (81) | 44.2 (52) | 20.7 (63) | 113 (37) | 108 (33)
  Week 2 | 0.000800 (173) | 0.181 (136) | 1.39 (116) | 1.97 (145) | 8.31 (77) | 55.1 (63) | 63.9 (46) | 194.8 (36)
  Week 3: number analyzed (Participants) | 3 | 6 | 2 | 17 | 14 | 6 | 5 | 6
  Week 3 | 0.000283 (145) | 0.460 (121) | 42.7 (73) | 4.18 (133) | 18.6 (71) | 75.9 (78) | 91.0 (52) | 347.3 (36)

9. Secondary Outcome: PK Assessment: Phase 1: Predicted Cumulative Area Under the Plasma Concentration Curve (AUC) of Isatuximab Over the First Week (0-168 Hours) (AUC1W)
Description: as for outcome 8
Time Frame: as for outcome 6
Population: Analysis was performed on PK population. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hour/mL
Arm/Group | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 3 | 6 | 3 | 18 | 16 | 6 | 6 | 7
mcg*hour/mL | 222 (80) | 2624 (24) | 7174 (54) | 11566 (48) | 13480 (38) | 12680 (35) | 32739 (28) | 28405 (27)

10. Secondary Outcome: PK Assessment: Phase 1: Predicted Cumulative Area Under the Plasma Concentration Curve (AUC) of Isatuximab Over the First 2 Weeks (0-336 Hours) (AUC2W)
Description: as for outcome 8
Time Frame: For Q2W:Cycle 1,Day 1: pre-dose, 15 min after start of infusion, at the end of infusion, 3, 7, 24, 48 and 336 hr post-infusion; For QW: Cycle 1,Day 1: pre-dose, 15 min after start of infusion, at the end of infusion, 4, 24, 48, 72 and 336 hr post-infusion
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hour/mL
Arm/Group | Phase 1: Isatuximab 1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 3 | 6 | 3 | 18 | 16 | 6 | 6 | 7
mcg*hour/mL | 222 (80) | 3076 (35) | 9546 (70) | 14876 (64) | 18967 (44) | 30187 (40) | 48003 (31) | 71174 (29)

11. Secondary Outcome: Pharmacodynamic (PD) Assessment: Phase 1: Change From Baseline in Serum/Plasma Markers
Description: Serum/plasma markers included: tumor necrosis factor alpha (TNF-α), interleukin-1β (IL-1-β), interleukin 6 (IL-6) and interferon-gamma (IFN-Gamma). Due to change in planned analysis, data for high-sensitivity C-reactive protein (hs-CRP) and CD38 was not collected and analyzed.
Time Frame: Cycle 1 Day 1
Population: Analysis was performed on all randomized participants who gave their informed consent, had received at least 1 dose (even incomplete) of isatuximab and had an assessable PD parameter. Here, 'number analyzed' = number of participants with available data for each category.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Groups:
- Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma): Participants with CD38+ HM along with participants with standard risk multiple myeloma , received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma): Participants with CD38+ HM along with participants with high risk multiple myeloma, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 10mg/kg QW: Participants with CD38+ HM, received Isatuximab 10 mg/kg, as IV infusion QW, i.e. on Day 1 and 8 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1:Isatuximab <=1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 16 | 6 | 3 | 26 | 18 | 6 | 7 | 7
picogram/milliliter (pg/mL)
  TNF alpha: number analyzed (Participants) | 16 | 5 | 3 | 23 | 16 | 6 | 6 | 5
  TNF alpha | 163.181 (253.373) | 179.783 (191.455) | 352.974 (220.394) | 340.799 (341.100) | 503.462 (479.813) | 342.664 (410.245) | 307.319 (398.025) | 412.541 (243.169)
  IL-1 Beta: number analyzed (Participants) | 15 | 4 | 3 | 21 | 16 | 6 | 6 | 5
  IL-1 Beta | 64.577 (227.399) | 29.741 (55.515) | 7.527 (8.118) | 299.058 (572.260) | 547.770 (1454.175) | 327.957 (759.305) | 305.914 (621.754) | 293.307 (612.746)
  IL-6: number analyzed (Participants) | 16 | 5 | 3 | 23 | 16 | 6 | 6 | 5
  IL-6 | 139.234 (212.385) | 261.732 (270.119) | 73.899 (53.211) | 148.594 (175.719) | 173.004 (433.297) | -8.109 (45.845) | 274.616 (234.752) | 165.295 (203.451)
  IFN Gamma: number analyzed (Participants) | 15 | 3 | 3 | 23 | 16 | 6 | 6 | 5
  IFN Gamma | 477.116 (1673.063) | 5.376 (9.312) | 25.806 (44.698) | 445.772 (1043.982) | 568.806 (1022.000) | 627.089 (1527.647) | 448.387 (569.499) | 1487.097 (2693.826)

12. Secondary Outcome: Immunogenicity Assessment: Phase 1: Number of Participants With Treatment-Emergent And Treatment-Boosted Anti-drug Antibodies (ADA) Response
Description: ADA response was categorized as: treatment induced and treatment boosted response. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period (defined as the time from the first isatuximab administration until end of Phase 1) in participants without preexisting ADA (defined as: ADA that were present in samples drawn before treatment), including participants without pre-treatment (before treatment) samples. Treatment boosted ADA was defined as pre-existing ADA that increased at least 2 titer steps between pre-treatment (before treatment) and post-treatment.
Time Frame: Up to 120 weeks
Population: Analysis was performed on ADA evaluable population which included all treated participants with at least one ADA assessment with a reportable result during the ADA on-study observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1:Isatuximab <=1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 16 | 6 | 3 | 26 | 18 | 6 | 6 | 7
Participants
  Treatment-induced ADA | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1
  Treatment boosted ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Clinical Assessment: Phase 1: Percentage of Participants With Overall Response and Clinical Benefit: Assessed Using European Society for Blood and Marrow Transplantation (EBMT) Criteria
Description: OR defined as participants with complete response (CR) or partial response (PR) as best overall response (BOR). Clinical benefit: participants with minimal response (MR) or better as BOR. BOR: best sequential response from start of treatment through the entire study excluding any time point following start of other treatment. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow aspirates, no increase in size or number of lytic bone lesions. PR: >=50% reduction of serum M-protein, reduction in 24 h urinary M-protein by >=90% or <200mg, >=50% reduction in size/number of soft tissue plasmacytomas, no increase in size or number of lytic bone lesions. MR: 25 to 49% reduction in serum M-protein, 50-89% reduction in 24h urine M-protein, 25-49% reduction in size of soft tissue plasmacytomas, no increase in size or number of lytic bone lesions.
Time Frame: From the date of randomization to the date of first documentation of progression or death (due to any cause) (maximum duration: 120 weeks)
Population: Analysis was performed on all-treated population. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1: Isatuximab 1mg/kg Q2W: Participants with CD38+ HM, received Isatuximab 1 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
Arm/Group | Phase 1: Isatuximab 1mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 3 | 5 | 3 | 25 | 18 | 6 | 7 | 7
percentage of participants
  OR | 33.3 | 0 | 33.3 | 28.0 | 16.7 | 33.3 | 14.3 | 28.6
  Clinical benefit | 33.3 | 20.0 | 33.3 | 28.0 | 27.8 | 33.3 | 28.6 | 42.9

14. Secondary Outcome: Clinical Assessment: Phase 1: Duration of Response (DOR)
Description: DOR: time from first response (PR or better) to first documented tumor progression/death. Progression as per EBMT: >25% increase in serum monoclonal paraprotein level, which must also be an absolute increase of >= 5 g/l: confirmed by >=1 repeated investigation; >25% increase in 24h urinary light chain excretion, which must also be an absolute increase of >=200 mg/24 h:confirmed by >=1 repeated investigation; >25% increase in plasma cells in a bone marrow aspirate/on trephine biopsy, which must also be an absolute increase of >= 10%; definite increase in size of existing bone lesions/soft tissue plasmacytomas; development of new bone lesions/soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11·5 mg/dl or 2·8 mmol/l) not attributable to any other cause. PR: >=50% reduction of serum M-protein, reduction in 24h urinary M-protein by >=90% or <200mg, >=50% reduction in size/number of soft tissue plasmacytomas, no increase in size/number of lytic bone lesions.
Time Frame: From the date of first response to the date of first documentation of progression or death (due to any cause) (maximum duration: 120 weeks)
Population: Analysis was performed only on subset of participants who had response in Phase 1 and not for the reporting group with no response.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Phase 1: Isatuximab 1mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 1 | 1 | 7 | 3 | 2 | 1 | 2
months | 20.21 | 7.16 | 5.76 (4.62) | 10.70 (11.25) | 14.31 (7.50) | 3.94 | 8.82 (7.83)

15. Secondary Outcome: Clinical Assessment: Phase 1: Time to First Response (TTR)
Description: TTR was defined as the time from first dose of isatuximab to first response (PR or better). PR: >=50% reduction of serum M-protein, reduction in 24 h urinary M-protein by >=90% or <200mg, >=50% reduction in size/number of soft tissue plasmacytomas, no increase in size or number of lytic bone lesions.
Time Frame: From the date of first dose administration to the date of first response or death (due to any cause) (maximum duration: 120 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Phase 1: Isatuximab 1mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW
Number analyzed (Participants) | 1 | 1 | 7 | 3 | 2 | 1 | 2
months | 0.95 | 6.41 | 2.52 (3.77) | 1.96 (1.72) | 1.38 (0.65) | 1.18 | 1.46 (0.77)

16. Secondary Outcome: Clinical Assessment: Phase 1: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) (Karnofsky Performance Status)-Shift From Baseline Value to Best Value During Treatment
Description: ECOG performance status was measured on a 4 point scale to assess participant's performance status. 0=Normal, fully functional; 1=Fatigue without significant decrease in daily activity; 2=Fatigue with significant impairment of daily activities or bed rest <50% of waking hours; 3=Bed rest/sitting >50% of waking hours; 4=Bedridden or unable to care for self, where lower score indicated good performance status. Number of participants with Baseline ECOG PS score and corresponding changes to the best values (categorized as: Baseline ECOG 1, During Treatment ECOG 0; Baseline ECOG 2, During Treatment ECOG 0; Baseline ECOG 2, During Treatment ECOG 1) are reported.
Time Frame: At baseline, during treatment (Day 1 up to 120 weeks)
Population: Analysis was performed on AT population. Data for this outcome measure was planned to be collected and analyzed for a combined arm of overall Phase 1 AT population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Isatuximab: All participants who were enrolled in Phase 1 and received Isatuximab.
Arm/Group | Phase 1: Isatuximab
Number analyzed (Participants) | 89
Participants
  Baseline ECOG 1, During Treatment ECOG 0 | 11
  Baseline ECOG 2, During Treatment ECOG 0 | 2
  Baseline ECOG 2, During Treatment ECOG 1 | 11

17. Secondary Outcome: Clinical Assessment: Phase 1: Number of Participants With Eastern Cooperative Oncology Group Performance Status (Karnofsky Performance Status)-Shift From Baseline Value to Worst Value During Treatment
Description: ECOG performance status was measured on a 4 point scale to assess participant's performance status. 0=Normal, fully functional; 1=Fatigue without significant decrease in daily activity; 2=Fatigue with significant impairment of daily activities or bed rest <50% of waking hours; 3=Bed rest/sitting>50% of waking hours; 4=Bedridden or unable to care for self, where higher score indicated worst performance status. Number of participants with Baseline ECOG PS score and corresponding changes to the worst values (categorized as: Baseline ECOG 0, During Treatment ECOG 1; Baseline ECOG 2, During Treatment ECOG 1; Baseline ECOG 0, During Treatment ECOG 2; Baseline ECOG 1, During Treatment ECOG 2; Baseline ECOG 0, During Treatment ECOG 3; Baseline ECOG 1, During Treatment ECOG 3; Baseline ECOG 2, During Treatment ECOG 3) are reported.
Time Frame: At baseline, during treatment (up to 120 weeks)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Isatuximab
Number analyzed (Participants) | 89
Participants
  Baseline ECOG 0, During Treatment ECOG 1 | 8
  Baseline ECOG 2, During Treatment ECOG 1 | 1
  Baseline ECOG 0, During Treatment ECOG 2 | 3
  Baseline ECOG 1, During Treatment ECOG 2 | 20
  Baseline ECOG 0, During Treatment ECOG 3 | 1
  Baseline ECOG 1, During Treatment ECOG 3 | 2
  Baseline ECOG 2, During Treatment ECOG 3 | 1

18. Secondary Outcome: Phase 2 Stage 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: as for outcome 2
Time Frame: From Baseline up to 30 days after the last dose (maximum duration: 414 weeks for Stage 1a and 92 weeks for Stage 1b)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W: Participants with multiple Myeloma received Isatuximab 3 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 23 | 24 | 25 | 25
Participants | 22 | 24 | 25 | 25

19. Secondary Outcome: Phase 2 Stage 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. TEAEs were defined as AEs that developed or worsened during the on-treatment period which was defined as the period from the time of first dose of study treatment until 30 days after the last dose of study treatment.
Time Frame: From Baseline up to 30 days after the last dose (maximum duration: 301 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 109 | 55
Participants | 101 | 51

20. Secondary Outcome: Phase 2 Stage 1: Duration of Response
Description: DOR:Time from date of 1st IAC determined response (>= PR) that was subsequently confirmed, to date of first IAC determined PD/death, whichever happened earlier. updated IMWG criteria- PR:>=50% decrease in difference between involved and uninvolved FLC levels in place of M-protein criteria or a >=50% reduction in plasma cells in place of M-protein if baseline was ≥30%. If present at baseline a >=50% reduction in size of soft tissue plasmacytomas; PD: Increase of 25% from lowest response value in any of following: Serum M-protein >=0.5 g/dL absolute increase and/or urine M-protein >=200 mg/24 hours absolute increase and/or >10 mg/dL absolute increase in difference between involved and uninvolved FLC levels, >=10% bone marrow plasma cells (PCs), development of new bone lesions/soft tissue plasmacytomas or definite increase in size of existing bone lesions/soft tissue plasmacytomas, development of hypercalcemia (corrected serum calcium >11·5 mg/dl) attributed to PC proliferation disorder.
Time Frame: From the date of first response until disease progression or death or data cut-off (maximum duration: 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: Analysis was performed only on subset of population who had response in Phase 2 stage 1.
Measure: Mean (Standard Deviation); unit: months
Groups:
- Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W: Participants with multiple Myeloma received Isatuximab 3 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion on Day 1 and Day 15 of each 28-day cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion Q2W, i.e. on Day 1 and Day 15 of Cycle 1 and 2 (each cycle 28 days), then every 4 weeks (Q4W), i.e. on Day 1 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 77 weeks).
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 1 | 7 | 5 | 6
months | 1.91 | 11.17 (5.77) | 7.31 (3.65) | 8.11 (2.33)

21. Secondary Outcome: Phase 2 Stage 2: Duration of Response
Description: DOR: Time from date of 1st IAC determined response (>= PR) that was subsequently confirmed, to date of 1st IAC determined PD or death, whichever happened earlier. As per updated IMWG criteria-PR: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. ≥50% decrease in difference between involved and uninvolved FLC levels in place of M-protein criteria or ≥50% reduction in plasma cells in place of M-protein if baseline was ≥30%. If present at baseline ≥50% reduction in size of soft tissue plasmacytomas; PD: Increase of >25% from lowest response value in any one of following: Serum M-component (absolute increase must be >0.5 g/dL)4 and/or Urine M-component (absolute increase must be >200 mg/24 h) and/or >10 mg/dL absolute increase in difference between involved and uninvolved FLC levels, >=10% bone marrow plasma cell, development of hypercalcemia (corrected serum calcium >11.5 mg/dL) attributed solely to plasma cell proliferative disorder.
Time Frame: From the date of first response until disease progression or death or data cut-off (maximum duration: 97 weeks)
Population: Analysis was performed only on subset of population who had response in Phase 2 stage 2.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 26 | 24
months | 8.6 (5.2) | 10.9 (4.6)

22. Secondary Outcome: Phase 2 Stage 1: Percentage of Participants With Clinical Benefit
Description: Clinical benefit: participants with sCR, CR, VGPR, PR or MR as per IMWG criteria, determined by IAC. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytomas,<5% PCs in bone marrow aspirates. sCR: CR + normal FLC ratio (0.26-1.65), absence of clonal cells in bone marrow biopsy. VGPR: serum & urine M-component detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-component plus urine M-component level <100mg/24hours; PR: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours, ≥50% decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria or a ≥50% reduction in plasma cells in place of M-protein if baseline was ≥30%. If present at baseline, ≥50% size reduction in soft tissue plasmacytomas. MR:>=25 but <49% reduction in serum M-protein, reduction in 24h urine M-protein by 50-89%, 25-49% size reduction in soft tissue plasmacytomas.
Time Frame: From the date of randomization to the date of first documentation of progression or death (maximum duration: 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: Analysis was performed on AT population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 23 | 24 | 25 | 25
percentage of participants | 4.3 | 41.7 | 32.0 | 36.0

23. Secondary Outcome: Phase 2 Stage 2: Percentage of Participants With Clinical Benefit
Description: Clinical benefit:participants with sCR, CR, VGPR, PR or MR, per IMWG criteria, determined by IAC. CR:negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytomas,<5% plasma cells in bone marrow aspirates,normal FLC ratio(0.26-1.65) in participants with only FLC disease.sCR:CR+normal FLC ratio, absence of clonal cells in bone marrow biopsy.VGPR:serum & urine M-component detectable by immunofixation, not on electrophoresis/,>=90% reduction in serum M-component plus urine M-component level <100mg/24h/,>=90% decrease in difference between involved and uninvolved FLC levels; PR:>=50% reduction of serum M-protein, reduction in 24h urinary M-protein by >=90%/<200mg/24h,>50% decrease in difference between involved and uninvolved FLC in place of M-protein criteria, >=50% reduction in size/number of soft tissue plasmacytomas. MR:>=25 but <49% reduction in serum M-protein,reduction in 24h urine M-protein by 50-89%, 25-49% reduction in size of soft tissue plasmacytomas
Time Frame: From the date of randomization to the date of first documentation of progression or death (maximum duration: 97 weeks )
Population: Analysis was performed on AT population.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 109 | 55
percentage of participants | 43.1 | 54.5

24. Secondary Outcome: Phase 2 Stage 1: Progression Free Survival (PFS)
Description: PFS was defined as the time interval from the date of first isatuximab administration to the date of the first IAC-confirmed disease progression (PD) or date of death due to any cause, whichever came first. As per IMWG criteria, PD: Increase of > 25% from lowest response value in any one or more of the following: Serum M-component and/or (the absolute increase must be > 0.5 g/dL), Urine M-component and/or (the absolute increase must be > 200 mg/24 h), > 10mg/dL decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria, >10% absolute percentage of bone marrow plasma cell, definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas, development of hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that attributed solely to the plasma cell proliferative disorder. Analysis was performed by Kaplan-Meier method.
Time Frame: From the date of the first dose administration until progression or death, whichever occurred first (maximum duration: 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: Analysis was performed on AT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 23 | 24 | 25 | 25
months | 2.1 [1.02 to 5.49] | 9.6 [2.23 to NA] — Upper limit of confidence interval was not estimable due to less number of participants with event. | 4.4 [1.84 to 5.82] | 3.6 [1.91 to 9.20]

25. Secondary Outcome: Phase 2 Stage 2: Progression Free Survival
Description: PFS was defined as the time interval from the date of first isatuximab administration to the date of the first IAC-confirmed disease progression or the date of death due to any cause, whichever came first. As per IMWG criteria, PD: Increase of >25% from lowest response value in any one of the following: Serum M-component (the absolute increase must be >0.5 g/dL)4 and/or Urine M-component (the absolute increase must be >200 mg/24 h) and/or >10 mg/dL decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria, ≥10% bone marrow plasma cell, development of hypercalcemia (corrected serum calcium >11.5 mg/dL) attributed solely to the plasma cell proliferative disorder. Analysis was performed by Kaplan-Meier method.
Time Frame: From the date of the first dose administration until progression or death, whichever occurred first (maximum duration: 97 weeks)
Population: Analysis was performed on AT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 109 | 55
months | 4.86 [3.877 to 7.688] | 10.15 [4.862 to 17.347]

26. Secondary Outcome: Phase 2 Stage 1: Overall Survival (OS)
Description: OS was defined as the time interval from the date of first Isatuximab administration to death from any cause. Analysis was performed by Kaplan-Meier method.
Time Frame: From the date of randomization to date of death from any cause (maximum duration 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: Analysis was performed on AT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 23 | 24 | 25 | 25
months | 15.277 [4.7310 to NA] — Upper limit of Confidence Interval (CI) was not estimable, due to less number of participants with event. | 18.628 [7.7536 to 20.1068] | NA [8.4435 to NA] — Median and upper limit of CI was not estimable, due to less number of participants with event. | NA [8.3450 to NA] — Median and upper limit of CI was not estimable, due to less number of participants with event.

27. Secondary Outcome: Phase 2 Stage 2: Overall Survival
Description: as for outcome 26
Time Frame: From the date of randomization to date of death from any cause (maximum duration: 97 weeks)
Population: Analysis was performed on AT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 109 | 55
months | 18.92 [13.602 to 23.064] | 17.25 [15.409 to NA] — Upper limit of CI was not estimable, due to less number of participants with event.

28. Secondary Outcome: Phase 2 Stage 1: Change From Baseline in Health Related Quality of Life (HRQL) European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scores: Global Health Status
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain) & other single items. For each item, high score = high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favorable outcome with a best quality of life for participant.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10 and End of Treatment (EOT: anytime up to 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: Analysis was performed on AT population. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure and 'number analyzed' = number of participants with available data for each category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 22 | 21 | 24 | 22
score on a scale
  Cycle 2 day 1: number analyzed (Participants) | 14 | 15 | 19 | 18
  Cycle 2 day 1 | -8.33 (20.15) | 2.22 (16.51) | -3.95 (20.67) | 0.00 (15.39)
  Cycle 3 day 1: number analyzed (Participants) | 7 | 11 | 14 | 12
  Cycle 3 day 1 | 0.00 (19.25) | -0.76 (16.44) | 6.55 (19.66) | -2.08 (15.54)
  Cycle 4 day 1: number analyzed (Participants) | 4 | 11 | 11 | 9
  Cycle 4 day 1 | 0.00 (24.53) | -5.30 (21.50) | 6.06 (21.11) | 7.41 (8.78)
  Cycle 5 day 1: number analyzed (Participants) | 4 | 12 | 9 | 5
  Cycle 5 day 1 | 0.00 (24.53) | 0.69 (15.27) | 6.48 (21.15) | 5.00 (4.56)
  Cycle 6 day 1: number analyzed (Participants) | 4 | 9 | 7 | 4
  Cycle 6 day 1 | 12.50 (14.43) | -10.19 (25.27) | 5.95 (13.36) | 10.42 (7.98)
  Cycle 7 day 1: number analyzed (Participants) | 2 | 7 | 4 | 5
  Cycle 7 day 1 | 12.50 (5.89) | -3.57 (15.85) | 8.33 (11.79) | 6.67 (6.97)
  Cycle 8 day 1: number analyzed (Participants) | 2 | 6 | 4 | 4
  Cycle 8 day 1 | 0.00 (35.36) | -11.11 (18.76) | 4.17 (15.96) | 6.25 (10.49)
  Cycle 9 day 1: number analyzed (Participants) | 2 | 5 | 4 | 4
  Cycle 9 day 1 | -8.33 (11.79) | -10.00 (19.90) | 4.17 (14.43) | 6.25 (10.49)
  Cycle 10 day 1: number analyzed (Participants) | 2 | 3 | 4 | 5
  Cycle 10 day 1 | -8.33 (35.36) | -16.67 (22.05) | 8.33 (11.79) | 3.33 (7.45)
  End of treatment: number analyzed (Participants) | 5 | 5 | 3 | 2
  End of treatment | 3.33 (33.64) | -11.67 (13.94) | -11.11 (20.97) | -12.50 (5.89)

29. Secondary Outcome: Phase 2 Stage 1: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Multiple Myeloma Specific Module With 20 Items (EORTC QLQ-MY20) Scores: Disease Symptom Subscale Score
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in participants with MM. It has 4 subscales: body image, future perspective), and 2 symptoms scales (disease symptoms and side-effects of treatment). Disease symptoms subscale used 4-point scale ranged from 1= 'Not at All' to 4= 'Very Much'. Scores were averaged, and transformed to 0 -100 scale, where higher scores = more symptoms and lower health-related quality of life (HRQL) and lower score = less symptoms and more HRQL.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10 and EOT (anytime up to 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 22 | 21 | 23 | 22
score on a scale
  Cycle 2 day 1: number analyzed (Participants) | 14 | 13 | 18 | 17
  Cycle 2 day 1 | 5.56 (18.36) | -3.42 (11.24) | 0.93 (13.91) | 2.61 (18.75)
  Cycle 3 day 1: number analyzed (Participants) | 7 | 11 | 13 | 11
  Cycle 3 day 1 | 7.94 (11.94) | -5.05 (14.15) | -5.98 (16.89) | -1.52 (13.17)
  Cycle 4 day 1: number analyzed (Participants) | 4 | 10 | 10 | 9
  Cycle 4 day 1 | 8.33 (13.22) | -3.89 (16.98) | -10.00 (16.93) | 0.62 (30.10)
  Cycle 5 day 1: number analyzed (Participants) | 4 | 11 | 8 | 5
  Cycle 5 day 1 | -6.94 (10.52) | 0.51 (19.95) | -9.03 (17.04) | -6.67 (17.74)
  Cycle 6 day 1: number analyzed (Participants) | 4 | 9 | 7 | 4
  Cycle 6 day 1 | 8.33 (7.17) | 1.23 (23.53) | -15.08 (20.96) | -6.94 (10.52)
  Cycle 7 day 1: number analyzed (Participants) | 2 | 6 | 4 | 5
  Cycle 7 day 1 | 2.78 (3.93) | -3.70 (22.95) | -18.06 (21.93) | -11.11 (11.79)
  Cycle 8 day 1: number analyzed (Participants) | 2 | 6 | 4 | 4
  Cycle 8 day 1 | -5.56 (7.86) | -2.78 (23.50) | -15.28 (23.30) | -4.17 (5.32)
  Cycle 9 day 1: number analyzed (Participants) | 2 | 5 | 4 | 4
  Cycle 9 day 1 | 5.56 (7.86) | -10.00 (10.69) | -16.67 (29.75) | -6.94 (12.32)
  Cycle 10 day 1: number analyzed (Participants) | 2 | 3 | 4 | 5
  Cycle 10 day 1 | 0.00 (0.00) | 0.00 (19.25) | -15.28 (30.56) | -6.67 (17.30)
  End of treatment: number analyzed (Participants) | 4 | 5 | 3 | 2
  End of treatment | -9.72 (19.44) | 7.78 (24.41) | 24.07 (22.45) | 25.00 (35.36)

30. Secondary Outcome: Phase 2 Stage 1: Change From Baseline in Euro Quality of Life 5 Dimension (EQ-5D) Generic Health Status - Visual Analogue Scale Scores
Description: EQ-5D was a standardized HRQL questionnaire consisting of EQ-5D descriptive system and Visual Analogue Scale (VAS). EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Day 1 of Cycles 4, 7, 10, 13, 16, 19, and EOT (anytime up to 77 weeks for Stage 1a arms and 53 weeks for stage 1b arm)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20mg/kg QW and Then Q2W
Number analyzed (Participants) | 22 | 21 | 22 | 22
score on a scale
  Cycle 4 day 1: number analyzed (Participants) | 4 | 9 | 9 | 9
  Cycle 4 day 1 | -5.75 (18.55) | 2.00 (16.88) | -4.78 (15.71) | 4.89 (16.02)
  Cycle 7 day 1: number analyzed (Participants) | 2 | 6 | 3 | 5
  Cycle 7 day 1 | -2.50 (0.71) | -6.00 (27.39) | 9.00 (18.25) | 1.00 (7.94)
  Cycle 10 day 1: number analyzed (Participants) | 2 | 3 | 3 | 5
  Cycle 10 day 1 | 0.50 (2.12) | -10.33 (9.29) | 10.33 (24.38) | -2.60 (8.11)
  Cycle 13 day 1: number analyzed (Participants) | 2 | 3 | 1 | 1
  Cycle 13 day 1 | 14.00 (19.80) | -5.00 (4.00) | -9.00 | -5.00
  Cycle 16 day 1: number analyzed (Participants) | 2 | 3 | 0 | 0
  Cycle 16 day 1 | 5.00 (5.66) | 0.67 (23.71) |  |
  Cycle 19 day 1: number analyzed (Participants) | 0 | 2 | 0 | 0
  Cycle 19 day 1 |  | -5.50 (4.95) |  |
  End of treatment: number analyzed (Participants) | 4 | 5 | 3 | 2
  End of treatment | -18.50 (16.98) | -11.60 (11.37) | -10.00 (9.54) | -9.00 (0.00)

31. Secondary Outcome: Pharmacokinetic Assessment: Phase 2 Stage 2: Area Under the Plasma Concentration Versus Time Curve of Isatuximab Over 1 Week Interval
Time Frame: Pre-dose, at the end of infusion, 1 hour and 168 hours post dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population which included participants who gave informed consent, received at least one dose (even if incomplete) of isatuximab, had an assessable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hour/mL
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 102 | 52
mcg*hour/mL | 37096 (80) | 35423 (88)

32. Secondary Outcome: Pharmacokinetic Assessment: Phase 2 Stage 2: Area Under the Plasma Concentration Versus Time Curve of Isatuximab Over 2 Weeks Interval
Time Frame: Cycle 1, Day 1: pre-dose, at the end of infusion, 168 and 336 hours post-infusion
Population: Analysis was performed on PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hour/mL
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 102 | 52
mcg*hour/mL | 91271 (78) | 86761 (77)

33. Secondary Outcome: Pharmacokinetic Assessment: Phase 2 Stage 2: Area Under the Plasma Concentration Versus Time Curve of Isatuximab Over 4 Weeks Interval
Time Frame: Cycle 1, Day 1: pre-dose, at the end of infusion, 168, 336, and 672 hours post-infusion
Population: Analysis was performed on PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hour/mL
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 102 | 52
mcg*hour/mL | 236360 (72) | 226372 (66)

34. Secondary Outcome: Pharmacokinetic Assessment: Phase 2 Stage 2: Plasma Concentration of Isatuximab Before Treatment Administration (Ctrough)
Time Frame: At Days 7, 14 and 28
Population: Analysis was performed on PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 102 | 52
mcg/mL
  Day 7 | 137 (75) | 128 (54)
  Day 14 | 230 (70) | 214 (57)
  Day 28 | 360 (63) | 305 (66)

35. Secondary Outcome: Pharmacokinetic Assessment: Phase 2 Stage 2: Accumulation Ratio of Isatuximab Based on Ctrough
Description: Ctrough is the plasma concentration observed before treatment administration. For 1st category, the accumulation ratio was calculated by dividing Ctrough value of Cycle 2 Day 1 by Cycle 1 Day 8 and for second category, accumulation ratio was calculated by dividing Ctrough value of Cycle 4 Day 1 by Cycle 1 Day 8.
Time Frame: Cycle 2, Day 1; Cycle 1, Day 8; Cycle 4, Day 1
Population: Analysis was performed on PK population. Here, 'number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 95 | 48
ratio
  Cycle 2 Day 1/Cycle 1 Day 8 | 521.38338 (4891.63390) | 3.24370 (1.73860)
  Cycle 4 Day 1/Cycle 1 Day 8 | 3.58378 (2.77398) | 3.95950 (3.19310)

36. Secondary Outcome: Immunogenicity Assessment: Phase 2 Stage 2: Number of Participants With Anti-drug Antibodies to Isatuximab
Description: ADA response was categorized as: treatment induced and treatment boosted response. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period (defined as the time from the first isatuximab administration until end of Phase 2 Stage 2) in participants without preexisting ADA (defined as: ADA that were present in samples drawn before treatment), including participants without pre-treatment (before treatment) samples. Treatment boosted ADA was defined as pre-existing ADA that increased at least 2 titer steps between pre-treatment (before treatment) and post-treatment.
Time Frame: Up to 97 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
Number analyzed (Participants) | 107 | 53
Participants
  Treatment induced ADA | 1 | 0
  Treatment boosted ADA | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signing of the informed consent form up to 30 days from last administration of study treatment (maximum exposure up to 120 weeks for Phase 1, 414 weeks for Phase 2 Stage 1a, 92 weeks for Phase 2 Stage 1b, and 301 weeks for Phase 2 Stage 2) regardless of seriousness or relationship to investigational product. All-cause mortality (Deaths) was collected for the entire study duration, 683 weeks
Description: Reported AEs were TEAEs which was defined as an AE that developed or worsened during the 'on treatment period' (time from the first dose of any study treatment up to 30 days after the last administration of the study treatment). Analysis was performed on AT population. For Phase 1, MedDRA 19.1 version was used and for Phase 2 Stage 1 and Phase 2 Stage 2, MedDRA 26.0 version was used.
Groups:
- Phase 1: Isatuximab <=1 mg/kg Q2W: Participants with CD38+ HM, received Isatuximab at any one of the dose <=1 mg/kg (i.e. either 0.0001 mg/kg or 0.001mg/kg or 0.01mg/kg or 0.03mg/kg, or 0.1mg/kg or 0.3 mg/kg or 1 mg/kg as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal by participant, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab 3mg/kg Q2W: Participants with CD38+HM, received Isatuximab 3 mg/kg, as IV infusion on Day 1 of each14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma): Participants with CD38+ HM along with participants with standard risk multiple myeloma were included this in arm and, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma): Participants with CD38+ HM along with participants with high risk multiple myeloma were included this in arm and, received Isatuximab 10 mg/kg, as IV infusion on Day 1 of each 14-day treatment cycle until occurrence of unacceptable toxicity, disease progression, death, consent withdrawal, investigator's decision, and/or availability of study drug (maximum exposure: 120 weeks).
- Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W: Participants with multiple Myeloma received Isatuximab 10 mg/kg, as IV infusion Q2W, i.e. on Day 1, 8, 15 and 22 of Cycle 1 and 2 (each cycle 28 days), then Q2W, i.e. on Day 1 and Day 15 of each 28-days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 414 weeks).
- Phase 2 Stage 1b: Isatuximab 20 mg/kg QW and Then Q2W: Participants with multiple Myeloma received Isatuximab 20 mg/kg, as IV infusion on Day 1 and Day 15 of Cycle 1 and 2 (each cycle 28 days), then Day 1 of each 28-days cycle until Unacceptable AE, disease progression, poor compliance to the study protocol, study termination or lost to follow up (maximum exposure: 92 weeks).
- Phase 2 Stage 2: Isatuximab Alone: Participants with relapsed or RRMM, received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 301 weeks).
- Phase 2 Stage 2: Isatuximab + Dexamethasone: Participants with relapsed or RRMM, received Isatuximab 20 mg/kg, as IV infusion on Day 1, 8, 15 and Day 22 of Cycle 1 (28 days) and then on Day 1 and 15 of each subsequent 28-day cycles along with dexamethasone: tablet or as IV infusion tablet or as IV infusion (40 mg/day for <75 years of age; 20 mg/day for >=75 years of age) on Days 1, 8, 15 and 22 of each 28 days cycle until unacceptable AE, disease progression, poor compliance to the study protocol, study termination, lost to follow up or investigator's decision (maximum exposure: 301 weeks).
Arm/Group | Phase 1: Isatuximab <=1 mg/kg Q2W | Phase 1: Isatuximab 3mg/kg Q2W | Phase 1: Isatuximab 5mg/kg Q2W | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) | Phase 1: Isatuximab 10mg/kg QW | Phase 1: Isatuximab 20mg/kg Q2W | Phase 1: Isatuximab 20mg/kg QW | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W | Phase 2 Stage 1b: Isatuximab 20 mg/kg QW and Then Q2W | Phase 2 Stage 2: Isatuximab Alone | Phase 2 Stage 2: Isatuximab + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 5/16 | 1/6 | 0/3 | 0/26 | 2/18 | 2/6 | 2/7 | 0/7 | 11/23 | 13/24 | 11/25 | 11/25 | 56/109 | 25/55
Serious Adverse Events (participants affected / at risk) | 3/16 | 3/6 | 1/3 | 10/26 | 10/18 | 3/6 | 3/7 | 3/7 | 13/23 | 11/24 | 10/25 | 9/25 | 52/109 | 27/55
Other Adverse Events (participants affected / at risk) | 16/16 | 6/6 | 3/3 | 26/26 | 18/18 | 6/6 | 6/7 | 6/7 | 22/23 | 23/24 | 25/25 | 24/25 | 92/109 | 47/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Isatuximab <=1 mg/kg Q2W (N=16) | Phase 1: Isatuximab 3mg/kg Q2W (N=6) | Phase 1: Isatuximab 5mg/kg Q2W (N=3) | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) (N=26) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) (N=18) | Phase 1: Isatuximab 10mg/kg QW (N=6) | Phase 1: Isatuximab 20mg/kg Q2W (N=7) | Phase 1: Isatuximab 20mg/kg QW (N=7) | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W (N=23) | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W (N=24) | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W (N=25) | Phase 2 Stage 1b: Isatuximab 20 mg/kg QW and Then Q2W (N=25) | Phase 2 Stage 2: Isatuximab Alone (N=109) | Phase 2 Stage 2: Isatuximab + Dexamethasone (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperviscosity Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia Of Malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Amyloidosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical Deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemophilus Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious Colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective Aortitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningococcal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 8 (10) | 5 (5)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonia Mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella Zoster Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma Of The Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 4 (4) | 3 (3)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea At Rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal Swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss Of Personal Independence In Daily Activities (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrinsic Iliac Vein Compression (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Isatuximab <=1 mg/kg Q2W (N=16) | Phase 1: Isatuximab 3mg/kg Q2W (N=6) | Phase 1: Isatuximab 5mg/kg Q2W (N=3) | Phase1:Isatuximab (CD38+HM and Standard Risk Multiple Myeloma) (N=26) | Phase 1: Isatuximab (CD38 + HM and High Risk Multiple Myeloma) (N=18) | Phase 1: Isatuximab 10mg/kg QW (N=6) | Phase 1: Isatuximab 20mg/kg Q2W (N=7) | Phase 1: Isatuximab 20mg/kg QW (N=7) | Phase 2 Stage 1a: Isatuximab 3mg/kg Q2W (N=23) | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W (N=24) | Phase 2 Stage 1a: Isatuximab 10mg/kg Q2W; Then Q4W (N=25) | Phase 2 Stage 1b: Isatuximab 20 mg/kg QW and Then Q2W (N=25) | Phase 2 Stage 2: Isatuximab Alone (N=109) | Phase 2 Stage 2: Isatuximab + Dexamethasone (N=55)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 0 (0) | 10 (13) | 4 (7) | 1 (2) | 0 (0) | 0 (0) | 9 (14) | 3 (3) | 8 (11) | 8 (12) | 4 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 5 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (9) | 3 (3) | 1 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Right Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 3 (3)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Scleral Discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 7 (8) | 1 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 4 (4) | 2 (3) | 2 (2) | 11 (13) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 6 (9) | 4 (6) | 1 (1) | 1 (1) | 2 (2) | 5 (7) | 7 (13) | 9 (11) | 5 (9) | 23 (37) | 11 (17)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2) | 1 (1) | 10 (13) | 6 (8) | 4 (6) | 1 (4) | 1 (1) | 6 (6) | 9 (14) | 11 (16) | 7 (8) | 16 (18) | 7 (32)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 6 (7) | 4 (5) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 4 (7) | 7 (9) | 6 (10) | 13 (15) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 8 (9) | 7 (7)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 6 (6) | 1 (1) | 2 (2)
Chills (General disorders) | 4 (6) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (5) | 5 (6) | 8 (12) | 2 (2) | 9 (10) | 4 (5)
Face Oedema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (10) | 2 (2) | 1 (1) | 8 (10) | 5 (6) | 4 (7) | 4 (6) | 1 (1) | 5 (5) | 7 (7) | 11 (12) | 9 (9) | 18 (106) | 11 (17)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 5 (6) | 1 (1) | 2 (3) | 5 (5) | 5 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 4 (5) | 5 (5) | 3 (3)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 1 (1) | 5 (6) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 5 (6) | 4 (4) | 3 (3) | 4 (4) | 7 (7)
Cytokine Release Syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular Cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 6 (8) | 2 (4)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (6) | 4 (5)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 4 (7) | 7 (8)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (5)
Tooth Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (4) | 1 (1) | 1 (1) | 7 (11) | 3 (3) | 3 (4) | 3 (4) | 1 (1) | 4 (5) | 7 (17) | 9 (20) | 6 (9) | 14 (16) | 8 (9)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 8 (9) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 2 (2) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 5 (7) | 3 (4) | 2 (2) | 12 (12) | 10 (13) | 4 (4) | 4 (4) | 3 (74) | 9 (11) | 13 (17) | 14 (14) | 15 (16) | 38 (41) | 20 (21)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scapula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Carbon Monoxide Diffusing Capacity Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T Wave Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Qrs Axis Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (4) | 3 (3) | 5 (5) | 11 (11) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (7) | 3 (5) | 5 (5) | 12 (15) | 5 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 7 (7) | 1 (2) | 0 (0) | 1 (5) | 2 (2) | 7 (8) | 3 (3) | 3 (3) | 20 (23) | 9 (10)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 10 (12) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 9 (9) | 5 (5)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 1 (1) | 8 (10) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (5) | 4 (4) | 8 (8) | 10 (13)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance Disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cranial Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Head Discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 2 (4) | 1 (33) | 4 (4) | 5 (6) | 7 (8) | 7 (8) | 15 (22) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Mental Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 5 (5)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vith Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Bradyphrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 2 (2) | 3 (3) | 2 (4) | 14 (19)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nipple Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 1 (1) | 6 (6) | 2 (3) | 3 (4) | 1 (1) | 2 (2) | 2 (3) | 10 (14) | 7 (10) | 8 (11) | 19 (22) | 12 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0) | 4 (5) | 5 (7) | 1 (2) | 3 (3) | 0 (0) | 5 (6) | 5 (6) | 8 (8) | 4 (4) | 17 (19) | 7 (7)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 6 (6) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 4 (5) | 3 (3) | 9 (10) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 3 (3) | 4 (4)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (2) | 5 (5) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 3 (3) | 1 (1) | 3 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 5 (5) | 3 (3)
Throat Lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (39) | 4 (4) | 1 (1) | 3 (4) | 4 (5) | 5 (5) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (8) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT01084252/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT01084252/SAP_003.pdf